CLINICAL TRIAL: NCT04304261
Title: Effects of Sodium-glucose Co-transporter-2 Inhibitors on the Cognitive Function in Type 2 Diabetic Patient
Brief Title: Effects of SGLT2i on the Cognitive Function in T2DM Patient (ESCDP)
Acronym: ESCDP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the Department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCDP
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2; Cognitive Functions Confusion
Keywords: Diabetes mellitus; Cognitive Functions; Sodium glucose transporter
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Confusion; Diabetes Mellitus | interventions — Canagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canagliflozin (Experimental): 12 weeks of Canagliflozin(100mg/day) treatment, randomly
  Interventions: Drug: Canagliflozin
- Sitagliptin (Experimental): 12 weeks of Sitagliptin (100mg/day) treatment, randomly
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Canagliflozin — 12 weeks of Canagliflozin(100mg/day) treatment
  Arms: Canagliflozin
Drug: Sitagliptin — 12 weeks of Sitagliptin (100mg/day) treatment
  Arms: Sitagliptin

SUMMARY:
Type 2 diabetes is associated with diabetic cognopathy, the prevalence of Alzheimer's Disease(AD) in T2DM patients is 1.5 to 2.5 times higher than the general population. Cognitive impairment seriously affects the health and quality of life of the elderly. Prevention and treatment measures for cognitive decline in persons with T2DM has not been well studied.

Sodium-glucose transporter-2 (SGLT-2) inhibitors, which lower serum glucose by inhibiting SGLT2-mediated glucose reabsorption in renal proximal tubules, could be neuroprotective. It was recently reported that the SGLT-2 inhibitor improved cognitive function and ameliorated oxidative stress via attenuating mitochondrial dysfunction, insulin resistance, inflammation, and apoptosis in mice or HFD-induced obese rats, that means SGLT-2 inhibitor may provide neuroprotection in the diabetic brain. Hence, Invokana (Canagliflozin) might act as a potent dual inhibitor of AChE and SGLT2. Since the development of diabetes is associated with AD, the design of new AChE inhibitors based on antidiabetic drug scaffolds would be particularly beneficial. Moreover, the present computational study reveals that Invokana (Canagliflozin) is expected to form the basis of a future dual therapy against diabetes associated neurological disorders.

The overall goal of this study is to explore the effects of SGLT2 inhibitor on the cognitive function in patients with type 2 diabetes mellitus and make further contribution to the improvement of cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Newly onset type 2 diabetes within 3 months
* 7%<HbA1c<10%

Exclusion Criteria:

* Type 2 diabetes with acute diabetic complications.
* Type1 diabetes.
* Thyroid dysfuncition.
* Any surgical or medical conditions that significantly influence absorption, distribution, metabolism or excretion of the intervention drugs.
* History of cardio-cerebral vascular events, such as congestive heart failure, myocardial infarction or stroke within 3 months.
* Hepatic insufficiency (AST or AST is twice higher than the upper limit) or history of hepatitis or cirrhosis, hepatic encephalopathy.
* Renal insufficiency (serum creatinine 1.5 times higher than the upper limit) or history of dialysis and nephritic syndrome.
* Acute infections, tumor, severe arrhythmia.
* Alcohol or medicine addiction, psychoactive substance abuse.
* Other diseases affecting cognitive function (congenital dementia, brain trauma, parkinson's diseases, toxicencephacopathy,epilepsy, mental disorders, severe lungdy sfunction, epilepsy, severe hypoglycemic coma, cerebrovascular disease, ischemic heart disease, etc.)
* Fertile woman without contraceptives.
* Allergic to or have contraindication to the intervention drugs.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Changes of cognitive function assessed by cognitive function scale | 12 weeks
  cognitive function scale

SECONDARY OUTCOMES:
Changes of standardized uptake values of brain and splanchnic organs assessed by 18F-PET-CT | 1 week
  18F-PET-CT
Changes of brain function assessed by near infrared brain functional imaging | 4 week
  near infrared brain functional imaging
Changes of urinary sodium and glucose excretion (mmol/24h) | 1 week
  urinary sodium and glucose excretion

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiming Zhu, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No